CLINICAL TRIAL: NCT04215380
Title: Effects of Gum Arabic Ingestion on Hormonal and Metabolic Changes in Patients With Polycystic Ovary Syndrome: Two Arm Randomized Double Blind Placebo Controlled Study
Brief Title: Effects of Gum Arabic Ingestion on Hormonal and Metabolic Changes in Patients With Polycystic Ovary Syndrome
Acronym: GA&PCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lamis Kaddam (Other)
Responsible Party: Sponsor-Investigator, Lamis Kaddam, Director, Al-Neelain University
Organization: Al-Neelain University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA& PCO
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Gum Arabic; Pectins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This arm will receive 100% natural Gum Arabic provided in a powder form as 30-grams-dose for 12 weeks
  Interventions: Dietary Supplement: Acacia Senegal extract
- Control group (Placebo Comparator): This group will be provided with pectin powder provided as two-gram-dose fo
  Interventions: Dietary Supplement: Pectin

INTERVENTIONS:
Dietary Supplement: Acacia Senegal extract — Oral Digestion of Gum Arabic dissolved in 200 ml of water to be consumed early morning in daily basis for 12 weeks
  Other Names: (Gum Arabic)
  Arms: Intervention Group
Dietary Supplement: Pectin — Oral Digestion of Pectin to be consumed early morning in daily basis for 12 weeks
  Arms: Control group

SUMMARY:
To assess the effects on hormonal and metabolic changes in the PCOs patients after ingestion of Arabic gum

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 5-20% of women of reproductive age worldwide it increases the risk for type 2 diabetes mellitus, cerebrovascular and cardiovascular events and not to mention it is one of the main causes of infertility. in the management of PCOS life style modification like weight reduction is necessary and recently it was discovered that GA ingestion causes significant reduction in BMI and body fat percentage among healthy adult females.so if GA could also affect the hormones and the metabolic changes in PCOs is going to be useful in decreasing the comorbidities and even treating PCOs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with PCO by independent Gynecologist

Exclusion Criteria:

* Diabetic patients
* Menopausal women
* History of allergy to Gum Arabic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2020-01-25 (Estimated); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
hormonal changes | 12 weeks
  Measure changes from the baseline values regarding LH, FSH, and testosterone level

SECONDARY OUTCOMES:
Metabolic change Serum cholestrol | 12 weeks
  Measure decrease from the baseline values regarding serum cholesterol level
Metabolic change HBA1C | 12 weeks
  Measure decrease from the baseline values regarding HBA1c
Body Mass index | 12 weeks
  Measure decrease from the baseline values regarding BMI

CONTACTS AND LOCATIONS:
Overall Officials: Imad M Fdl-Elmula, PhD, Study Director — Alneelain University
Locations (1):
- Banoon center for assisted reproduction and, obstetrics and gynecology, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, CSR

REFERENCES:
- [Background] Babiker R, Elmusharaf K, Keogh MB, Saeed AM. Effect of Gum Arabic (Acacia Senegal) supplementation on visceral adiposity index (VAI) and blood pressure in patients with type 2 diabetes mellitus as indicators of cardiovascular disease (CVD): a randomized and placebo-controlled clinical trial. Lipids Health Dis. 2018 Mar 20;17(1):56. doi: 10.1186/s12944-018-0711-y. PMID 29558953
- [Background] Esmaeilzadeh S, Andarieh MG, Ghadimi R, Delavar MA. Body mass index and gonadotropin hormones (LH & FSH) associate with clinical symptoms among women with polycystic ovary syndrome. Glob J Health Sci. 2014 Sep 28;7(2):101-6. doi: 10.5539/gjhs.v7n2p101. PMID 25716399
- [Background] Kaddam L, Fadl-Elmula I, Eisawi OA, Abdelrazig HA, Saeed AM. Acacia Senegal (Gum Arabic) Supplementation Modulate Lipid Profile and Ameliorated Dyslipidemia among Sickle Cell Anemia Patients. J Lipids. 2019 Jun 18;2019:3129461. doi: 10.1155/2019/3129461. eCollection 2019. PMID 31316836